CLINICAL TRIAL: NCT05959759
Title: Dimethyl Fumarate Treatment for Intracranial Unruptured Aneurysms: a Double Blind Randomized Controlled Trail
Brief Title: Dimethyl Fumarate Treatment for Intracranial Unruptured Aneurysms.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other); Beijing Chao Yang Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTHDMF
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Intracranial Aneurysm; Aneurysm, Brain; Inflammation Vascular
Keywords: Dimethyl Fumarate; High resolution magnetic resonance
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Dimethyl Fumarate

STUDY DESIGN:
Intervention Model Description: A total of 60 patients will be enrolled in this study. Randomly divide the patients into experimental group and placebo group according to 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients with intracranial aneurysms will be numbered and randomly divided into two groups, 30 patients in each group, and seal them. Through blind method, one group will be given dimethyl fumarate enteric capsule (the initial dose is 120 mg twice a day, and after 7 days, the dose will be increased to the maintenance dose of 240 mg twice a day, for 6 months). The other group took placebo with the same appearance (color, taste, size, shape) as the test drug.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dimethyl fumarate (Experimental): dimethyl fumarate enteric capsule (the initial dose is 120 mg twice a day, and after 7 days, the dose will be increased to the maintenance dose of 240 mg twice a day, for 6 months)
  Interventions: Drug: Dimethyl fumarate
- Placebo (Placebo Comparator): placebo with the same appearance (color, taste, size, shape)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl fumarate — dimethyl fumarate enteric capsule (the initial dose is 120 mg twice a day, and after 7 days, the dose will be increased to the maintenance dose of 240 mg twice a day, for 6 months), 30 patients for this arm.
  Arms: Dimethyl fumarate
Drug: Placebo — placebo with the same appearance (color, taste, size, shape), 30 patients for this arm.
  Arms: Placebo

SUMMARY:
This study was designed to identify whether there is a measurable reduction in inflammation in walls of intracranial aneurysms with oral dimethyl fumarate.

DETAILED DESCRIPTION:
Intracranial aneurysm (IA) is a common cerebrovascular disease and the main cause of nontraumatic subarachnoid hemorrhage. Once ruptured, it will cause a high mortality rate, and nearly half of the survivors will also have disabilities. After comparing surgical risk and rupture risk, a significant proportion of patients with intracranial aneurysms choose conservative observation.

Previous studies suggest that inflammation of aneurysmal wall is a high-risk factor of rupture. Dimethyl fumarate (DMF) acts as an anti-inflammatory agent by activating nuclear factor erythroid 2-related factor 2(Nrf2) and other pathways. Animal experiments found dimethyl fumarate reduces the formation and rupture of intracranial aneurysms.

MRI High-resolution vessel wall imaging (HR-VWI) has become a valuable method to assess the Wall of unruptured intracranial aneurysms. Using HR-VWI, it may be possible to detect smaller or more subtle areas of signal enhancement and change, which may give a more precise understanding of the pathology.

In this study, DMF was evaluated for its ability to reduce inflammation of the aneurysm wall measured with High-resolution Vessel Wall Imaging (HR-VWI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years.
2. Unruptured IA of ≥3mm identified on imaging (CT, MRI or digital subtraction angiography).
3. Aneurysm wall enhancement identified by HR-VWI before treatment.
4. Ability to understand the objective of the trial with provision of written informed consent.

Exclusion Criteria:

1. MRI contraindications (metallic implant, contrast allergy, claustrophobia, etc).
2. Planned treatment of the aneurysm within 12 months.
3. Current treatment with drugs that might have an anti-inflammatory effect (aspirin, statins, immunosuppressive drugs, etc.).
4. Severely impaired liver or renal function.
5. Retreatment of recurrent aneurysm.
6. Pregnant or lactating women.
7. Malignant diseases (liver disease, kidney disease, congestive heart failure, malignant tumours, etc.).
8. Poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of aneurysm wall inflammation as measured by HR-VW-MRI. | 6 months
  Change of aneurysm wall enhancement index of at least 20% on HR-VM-MRI at the end of 6 months of dimethyl fumarate treatment, compared to no treatment.

SECONDARY OUTCOMES:
Change of aneurysmal morphology parameter | 6 months
  The proportion of morphological growth of aneurysms from before treatment to the 6 months follow-up. An increase ≥ 1mm in any diameter or the appearance of a daughter sac will be defined as growth in aneurysmal morphology.
Change of inflammatory markers in patients | 6 months
  Changes in CRP, TNF-α, IL-1β and IL-6 in patients with unruptured IAs from before treatment to the 6 months follow-up. The CRP, TNF-α, IL-1β and IL-6 levels will be measured at before treatment and at 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yisen Zhang, MD, Study Director — Beijing Neurosurgical Institute & Beijing Tiantan Hospital
Locations (1):
- Beijing Neurosurgical Institute & Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data are available on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: Data are available on reasonable request.

REFERENCES:
- [Derived] Huang J, Zhang Y, Turhon M, Zheng Z, Li W, Kang H, Wang C, Liu J, Jiang P. Dimethyl fumarate treatment for unruptured intracranial aneurysms: a study protocol for a double-blind randomised controlled trial. BMJ Open. 2024 May 21;14(5):e080333. doi: 10.1136/bmjopen-2023-080333. PMID 38772883